CLINICAL TRIAL: NCT04964687
Title: Impact of Integrating an Addiction Team on Post Liver Transplantation Survival for Alcohol-related Liver Disease and Its Complications: a Multicenter Retrospective Comparative Study.
Brief Title: Impact of Integrating an Addiction Team on Post Liver Transplantation Survival for Alcohol-related Liver Disease and Its Complications.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0410
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Alcoholism; Alcohol Use Disorder; Alcohol; Liver
Keywords: transplantation liver; hepatocellular carcinoma; Alcohol
MeSH Terms: conditions — Alcoholism; Liver Diseases, Alcoholic; Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transplanted patients seen by an addictionology team: Adult patients with alcohol-related liver disease, possibly complicated by hepatocellular carcinoma, that required liver transplantation in participating centers from January 2000 to December 2015, and seen by an addictology team before and after the transplantation.
  Interventions: Procedure: Liver transplantation
- Transplanted patients not seen by an addictionology team: Adult patients with alcohol-related liver disease, possibly complicated by hepatocellular carcinoma, that required liver transplantation in participating centers from January 2000 to December 2015, and seen by an addictology team before and after the transplantation.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation

SUMMARY:
Investigator seeks to determine wether integrating an addiction team into a liver transplantation unit improves the prognosis of patients with alcohol-related liver disease requiring liver transplantation. Our hypothesis is that patients managed by an addiction team before and after liver transplantation have less frequent alcohol relapses, thus decreasing the risk of cardiovascular complications, de novo cancer, recurrence of alcohol-related cirrhosis, and consequently increasing their overall survival.

DETAILED DESCRIPTION:
In this observational, retrospective and multicentre study, investigator seek to determine the effect of integrating an addiction team into liver transplantation unit on prognosis of patients with alcohol-related liver disease requiring liver transplantation. Investigatore plan to compare patients in 2 groups, depending on whether they have received or not specific addiction care before and after transplantation. This study was conducted over a period of 15 years in three French liver transplant units.

ELIGIBILITY:
Inclusion criteria:

* adult patients
* who received a liver transplant between January 2000 and December 2015 for alcohol-related liver disease as a primary or secondary indication (hepatocellular carcinoma)
* who survived for more than 6 months after their liver transplant.

Exclusion criteria:

* association of other causes of hepatopathy: viral hepatitis B or C, hereditary hemochromatosis.
* death before discharge from hospital after liver transplantation.
* patient unwilling to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with alcohol-related liver disease, possibly complicated by hepatocellular carcinoma, that required liver transplantation in participating centers from January 2000 to December 2015.
  * Saint Eloi University Hospital, University of Montpellier
  * Edouard Herriot University Hospital, Hospices Civils de Lyon
  * Rangueil University Hospital, University of Toulouse
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients transplanted for alcoholic liver disease. | Date of last news (at least 5 years for surviving patients)
  Patient time (delay between date of transplantation and date of last news) + state (alive or deceased)

SECONDARY OUTCOMES:
Alcohol relapse rate | Date of last news (at least 5 years for surviving)
  Number of patients with alcohol relapse among all transplanted patients.
Severe alcohol relapse rate | Date of last news (at least 5 years for surviving)
  Number of patients with severe alcohol relapse among all transplanted patients
Rate of alcohol-related cirrhosis recurrence | Date of last news (at least 5 years for surviving)
  Number of patients with alcohol-related cirrhosis among all transplanted patients.
Rate of development of cardiovascular risk factors | Date of last news (at least 5 years for surviving)
  Number of patients developing one or more cardiovascular risk factors (hypertension, dyslipidemia, diabetes, smoking) among all transplanted patients.
Cardiovascular event rate | Date of last news (at least 5 years for surviving)
  Number of patients with one or more cardiovascular events (coronary syndrome, stroke, arterial disease) among all transplant patients.
De novo cancer-free survival | Date of last news (at least 5 years for surviving)
  Number of patients developing de novo cancer as a function of time among all transplanted patients

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu-Rigole, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Daniel J, Dumortier J, Del Bello A, Gamon L, Molinari N, Faure S, Meszaros M, Ursic-Bedoya J, Meunier L, Monet C, Navarro F, Boillot O, Pageaux GP, Donnadieu-Rigole H. Integrating an addiction team into the management of patients transplanted for alcohol-associated liver disease reduces the risk of severe relapse. JHEP Rep. 2023 Jul 30;5(10):100832. doi: 10.1016/j.jhepr.2023.100832. eCollection 2023 Oct. PMID 37681206